CLINICAL TRIAL: NCT04725747
Title: A Randomized, Double-Masked, Controlled, Single Site Investigator Initiated, Exploratory Study of the Midazolam/Ketamine Melt vs Ketamine Melt Alone vs Midazolam Melt Alone in Subjects Undergoing Intraocular Surgery.
Acronym: MAKER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Principal Investigator, John Berdahl, MD, MD, Vance Thompson Vision
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAKER
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Midazolam; Ketamine; Administration, Sublingual

STUDY DESIGN:
Intervention Model Description: 1:1:1 treatment arms. Arm 1 Ketamine/Midazolam melt. Arm 2 Ketamine melt. Arm 3 Midazolam melt.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double masked study in which the doctor/nurse anesthetist evaluating the subject with the Ramsey scale will be masked to the treatment given. The subject will also be masked to the treatment group and the study/control drug.
  To keep the doctor/nurse anesthetist masked, the unmasked nurse will prepare the study/control drug and then administer it to the subject without unmasking the doctor/nurse anesthetist or the subject. The unmasked nurse will administer one 3/50mg MK melt, or one 3mg Midazolam melt, or one 50mg Ketamine melt sublingually based on the subject's randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Midazolam/Ketamine Melt (Experimental): One Midazolam/Ketamine 3mg/50mg melt administered sublingually
  Interventions: Drug: Midazolam/Ketamine HCl 3mg-50mg sublingual
- Midazolam Melt (Active Comparator): Midazolam 3mg melt administered sublingually
  Interventions: Drug: Midazolam 3mg Sublingual
- Ketamine Melt (Active Comparator): Ketamine 50mg melt administered sublingually
  Interventions: Drug: Ketamine 50mg Sublingual

INTERVENTIONS:
Drug: Midazolam/Ketamine HCl 3mg-50mg sublingual — Single sublingual administration of Midazolam/Ketamine HCl 3mg-50mg sublingually prior to surgery
  Arms: Midazolam/Ketamine Melt
Drug: Midazolam 3mg Sublingual — Single sublingual administration of Midazolam 3mg sublingually prior to surgery
  Arms: Midazolam Melt
Drug: Ketamine 50mg Sublingual — Single sublingual administration of Ketamine HCl 50mg sublingually prior to surgery
  Arms: Ketamine Melt

SUMMARY:
This study is designed to explore the sedative and analgesic effectiveness of the Midazolam/Ketamine melt compared to Midazolam melt alone or Ketamine melt alone in subjects undergoing intraocular surgery.

DETAILED DESCRIPTION:
Cataract surgery today is a highly effective and efficient procedure, with average times for completion ranging around 15 minutes in duration. Patients undergoing cataract surgery are typically given sedatives and often times pain medication (e.g. opioids) just prior to and during the procedure. The overwhelming majority of patients are given these medications via intravenous administration. The insertion of an IV line has been associated with patient complaints of pain and bruising, and can increase the administrative burden on the clinical staff. In addition to the national crisis surrounding opioid abuse, opioids have many negative side effects during cataract surgery such as respiratory depression, dizziness, nausea, and post- operative vomiting.

To reduce the side effects, improve patient satisfaction, and help surgical center flow the Midazolam/Ketamine melt (MK Melt) has been suggested as an alternative to provide sedation and analgesia in subjects undergoing minor outpatient surgery, such as cataract surgery. The addition of ketamine should provide enough analgesia for the mild discomfort reported during cataract surgery. This study is intended to evaluate the MK Melt and its ability to provide an adequate level of both sedation and intraoperative pain control vs an active control.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male or female, and between the ages of 55-80 years old.
2. Subjects willing and able to sign the informed consent and capable of committing to the duration of the study.
3. Subjects undergoing uncomplicated stand-alone cataract surgery without planned use of Omidria or intra-operative lidocaine.
4. Subjects that are willing to have an IV placed prior to intraocular surgery
5. Subjects undergoing first eye cataract surgery
6. Subjects that in the opinion of the investigator can tolerate 1 dose of MK 3/50 Melt.

Exclusion Criteria:

1. Subjects who have undergone sedation in the past 90 days.
2. Women who are pregnant or lactating at the time of the study.
3. Subjects who do not wish to or cannot comply with study procedures.
4. Subject with any cognitive impairment (i.e: Alzheimer's, dementia, etc.) that in the opinion of the investigator may confound the study results.
5. Subjects with history of substance abuse.
6. Subjects that are currently taking a prescription pain medication.
7. Subjects that are not willing to abstain from all over-the-counter pain medication with the exception of 500-1000mg acetaminophen for 24 hours prior to surgery.
8. Subjects that are not willing to abstain from NSAID or steroid eye drops prior to surgery.
9. Subjects with planned use of femtosecond laser, zepto, iris hooks or a malyugin ring during cataract surgery.
10. Subjects with chronic pain rated moderate to severe within the past week.
11. Subjects that have a psychiatric disorder that is currently uncontrolled.
12. Subjects scheduled for same day bilateral or second eye cataract surgery.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of Sedation | Duration of surgery
  The Doctor/Nurse Anesthetist will evaluate the subject's level of sedation on the
  Ramsey Sedation Scale. Adequate sedation demonstrated by a score of 2 or higher on the Ramsey Scale:
  * Upon entering operative room (before being prepped and draped)
  * Immediately post-op upon entering the PACU
  The Ramsey scale is:
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response
  Source: Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxolone-alphadalone. BMJ. 1974;2:656-659.
Level of Pain | Duration of surgery
  Adequate pain control demonstrated by a score of 3 or below on the Numeric Pain Rating Scale (NPRS) by asking the following questions at the following times:
  1. "How painful was that on a scale of 0=no pain to 10=extreme pain?" will be asked:
     * Upon insertion of the speculum
     * Upon first incision
     * Upon insertion of phacoemulsification probe
     * Upon Lens insertion
     * Upon removal of sterile drape
  2. "How would you rate your worst pain during surgery on a scale of 0=no pain to 10=extreme pain?" will be asked:
     * Immediately after surgery in the OR
     * 10-15 mins after the subject reaches the PACU
  3. "On a scale of 0=no pain to 10=extreme pain what number best describes your overall pain during the surgery?" Will be asked:
     * Immediately after surgery in the OR
     * 10-15 mins after the subject reaches the PACU
Need for Rescue Medication | Duration of surgery
  Percentage of patients requiring rescue medication (IV Fentanyl) for pain. Rescue medication will only be giving if a subject reports a pain level of 4 or higher on the NPRS.

SECONDARY OUTCOMES:
Eye Movement During Surgery | Duration of surgery
  Eye movement during surgery (evaluated by a masked evaluator by reviewing operative recording).
Clinician's Global Impression | Duration of surgery
  Clinician's impression of patient's sedation during surgery
Patient Satisfaction | 1 day post operatively
  Patient satisfactions, determined by asking the patient "How satisfied were you with your overall experience?" at the one-day post-op or via phone call one-day post-op.

OTHER OUTCOMES:
Blood pressure changes | Duration of surgery
  Blood pressure will be tracked at 3-5 minute intervals throughout the surgery. Any changes in blood pressure >20mmHg in systolic or diastolic will be identified as a clinically meaningful change.
Heart rate changes | Duration of surgery
  Heart rate will be tracked at 3-5 minute intervals throughout the surgery. Any changes in heart rates greater than 100 beats per minute or less than 60 beats per minute will be identified as a clinically meaningful change.

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No